CLINICAL TRIAL: NCT05229302
Title: Testing the Effectiveness of a CBT Online-based Program to Reduce Suicide Ideation Among School Adolescents in Chile: A Cluster Randomized Controlled Trial
Brief Title: Effectiveness of a CBT Online-based Program to Reduce Suicide Ideation Among School Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Talca (Other)
Collaborators: Universidad de los Andes, Chile (Other); Centre for Youth Mental Health, University of Melbourne, Australia (Unknown)
Responsible Party: Principal Investigator, Daniel Nunez, Associate Professor, University of Talca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Fondecyt_1210093
Record Dates: First submitted 2021-11-29; First posted 2022-02-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Suicidal Ideation
Keywords: Suicidal ideation; Web-based intervention; Effectiveness; Adolescents
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The Outcome Assessor will be unaware of which treatment arms participants have been assigned to El evaluador será ciego a la pertenencia de los participantes al grupo control o de intervención
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Secondary students with suicidal ideation participating in the intervention (Reframe-IT). The students will be referred to Primary care where they will be assessed by a physician who will determine if the adolescent could enter into the National Depression Treatment Program for people aged 15 and above, which is organized as a step care treatment
  Interventions: Behavioral: Reframet IT; Behavioral: Usual care
- Control (Active Comparator): Secondary students referred to Primary care where they will be assessed by a physician who will determine if the adolescent could enter into the National Depression Treatment Program for people aged 15 and above, which is organized as a step care treatment.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Reframet IT — The online intervention comprises 8 modules of cognitive behavioral therapy (CBT) delivered at schools by psychologists over 10 weeks. Contents: engagement and problem identification, emotional recognition and distress tolerance, identification of negative automatic thinking, help seeking and activity scheduling, problem solving, and cognitive restructuring, and a wrap up session. Two activities per module. Using a message board, the participant could communicate with research therapists who also check completed activities and respond with personalized messages. The face-to-face intervention comprises 4 CBT-based sessions to help the students in three aspects: i) close support and monitoring in case of an increase of symptomatology; ii) motivation to persist with the CBT; and iii) support the interaction between the students and CBT. Additionally, participants will be referred to a primary care clinic to receive treatment as usual.
  Arms: Intervention
Behavioral: Usual care — Treatment as usual consists of identification and assisted referral to a primary care clinic where trained psychologists will assess the symptomatology and propose a course of actions, from initiation of psychotherapy to referral to a General practitioner to initiate medication if needed. Psychoterapy in primary care clinics consists of a range of 4-8 sessions twice a month. Most of the content of the psychotherapy are based on Cognitive-Behavioral Model. When needed, general practioners may suggest using medication, which normally are SSRI anditepressant (e.g., Fluoxetine, Sertraline). Medical check-up is conducted every month or every two months.

SUMMARY:
This is a single-blind two armed cluster randomized controlled trial (cRCT) aimed to determine the effectiveness of an integrated blended intervention (online a face-to face sessions) to reduce suicidal ideation (primary outcome). Additionally, the effect of the program on the following secondary outcomes will be assessed: suicidal attempts, depressive symptoms, hopelessness and problem-solving skills. On the other side, given its probable role as underlying mechanism in SI reduction, the effect of the intervention on emotional regulation will be assessed. Moreover, the study will evaluate whether the effects of the cRCT on primary and secondary outcomes remain at post-intervention and at 3-month, 6-month and 12-month follow-up.

DETAILED DESCRIPTION:
1. Study design. This is a single-blind, two-armed randomized controlled trial evaluating changes in primary and secondary outcomes post-intervention and follow-up. The two arms will be: 1) The intervention, which comprises eight internet-based modules of CBT delivered over 10-week, and four 45-min face-to-face psychotherapeutic CBT sessions; and 2) Control group (Treatment-As-Usual).
2. Participants. Schools with secondary education (Grades 9-12), mixed-sex, located in three different cities in the South of Chile (Talca, Linares, Curicó) with three classes per year.
3. Sample size. It is expected to recruit at least ten schools per arm, allocated on a 1:1 ratio. Each arm should include 140 eligible students. This sample size takes into account a loss at follow-up of 20% of the students. Considering a 20% of school rejection at the recruitment stage, it is expected to recruit 12 schools. Studies of similar school-based interventions report effect sizes of at least 0.4 standard deviation using symptoms questionnaires as proposed here. The results previously observed by Hetrick and colleagues and the clustersampsi command in Stata Software will be used to estimate the number of clusters in two arms, using the following command: clustersampsi, samplesize mu1(X1) mu2(X2) sd1(Y1) sd2(Y27) m(Z) rho(R). Where X1 = mean in arm 1; X2 = mean in arm 2; Y1 = standard deviation (SD) in arm 1; Y2 = SD in arm 2; Z = number of children per school on average (harmonic mean) (n = 14); and R = intracluster correlation. The two arms will be balanced for school size.
4. Process

   4.1. Recruitment. The potential participants will be schools with secondary education from three cities in Chile. The schools will learn about the study through invitations that will be made to their institutional email and social networks. Eligible schools will be invited through letters sent to the authorities who will sing a letter to participate in the study.

   4.1.1 Enrollment Strategy. This research project will be disseminated after the approval of the Scientific Ethics Committee. At the beginning of the academic year, a letter with information about the study and the written consent will be sent to all parents or main caregivers. To select the participants, all students attending to 9-12 Grades will be invited to participate in the study, and the students will be asked for a written assent. All consented/assented students will be surveyed with screening questionnaires during the second month of the academic year (C-SSRS, PHQ-9; CAPE-P-15). All students attending 9-12 grades in selected secondary schools and scoring > 3 points in the Columbia Severity Raging Scale (CSSR-S) will be invited to participate in the study. From previous data, it is expected to find 10% of students with suicidal thoughts. Students with intellectual disabilities and communication difficulties due to language will be excluded. Students with one or more suicide attempts during the last month (>11 on the PHQ-9 scale) and students with psychotic symptoms (>1.50 in the CAPE-P-15) will be also excluded. These students will be referred to Primary Care Centers and will be invited to use the intervention "Take care of your mood" ("Cuida Tu Ánimo; a universal intervention that shows beneficial effects for the prevention of depressive symptoms) available for free at the following link (http://cuidatuanimo.net), where students will find helpful information to prevent depressive symptoms. This intervention has been developed by a research team with whom Dr. Daniel Nunez collaborates.

   4.1.2. Informed consent will be requested from students. The students of the selected schools will be invited to participate in informative talks about the study. Once the study, inclusion and exclusion criteria have been explained, a description of the screening instruments, their importance, and the selection process will be provided to interested parties. The informed consent will be sent to those accepting participate by emails and signed digitally through Qualtrics. Qualtrics is a platform that allows information to be collected online, with high-security standards, and that also can facilitate the digital signature through a cell phone or tablet (using the finger) or through a computer (with a mouse). This platform will collect data of screening instruments: suicidal ideation (SI) and suicide attempts, depressive symptoms, and psychotic symptoms. These data will be used for the study eligibility analysis. All who report any level of SI during the previous month (score > 3 in the C-SSR) will be invited to participate in the following step of the study.

   Informed consent will cover both general screening and baseline measurements and follow-up during and after the intervention.

   4.2. Evaluation procedure. Self-report questionnaires assessing primary and secondary outcomes (SIQ; BDI-II; BHS, STAI-X, SPSI-R, ERQ-CA, CBTS), will be administered at baseline (one week before the start of the intervention), at post-intervention, and follow-up (3, 6 and 12 months).

   4.3. Randomization. Randomization will be performed once all schools are recruited. Schools will be randomly assigned to either group with a 1:1 allocation as per computer-generated randomization. An independent statistician will perform the randomization. Each arm should include 140 eligible students. This sample size takes into account a loss at follow-up of 20% of the students. Considering a 20% of school rejection at the recruitment stage, it is expected to recruit 12 schools. The two arms will be balanced for school size.

   4.4. Blind condition: By the nature of the intervention, the participants are not blind with respect to the group allocation (intervention or control group). The evaluations will be carried out through self-report questionnaires sent in electronic format, and their evaluation will be automatic, without human action. In data analysis, the statistician will be blind to the intervention group of participants.
5. Study duration. From its recruitment and enrollment phase to the last evaluations (follow-up), the entire study will last approximately 18 months.

   Participants will be enrolled once accept and consent to participate in the study. Once enrolled, the intervention will begin the following week to reduce, as much as possible, the possibility of variation in the results of their initial measurements between the previous evaluation period and the beginning of the intervention.
6. Intervention. The internet-based component: The intervention has been described elsewhere (Robinson et al., 2015; Hetrick et al., 2017). It comprises eight modules of CBT delivered over a 10-week intervention period. Each participant can access to a personalized web page accessed via secure login. The program will be administered at schools by trained school psychologists (1 psychologist per school). The authors will deliver the training of the program. Once each module was completed in the psychologist's presence, participants can access it from home, 24 hours a day. For safety reasons, the program does not have social networking functions. Standard CBT approaches are delivered in the intervention, with a specific focus on SI and behaviors. The topics covered by the eight modules are: engagement and problem identification, emotional recognition and distress tolerance, identification of automatic negative thinking, behavioral activation-help seeking, behavioral activation-activity scheduling (including relaxation techniques), problem-solving, and cognitive restructuring and a wrap-up session. This content is delivered via a series of video diaries by young people as main characters, with an adult 'host' character highlighting the CBT contents that had been presented in the context of the video diaries. There are two activities per module. The site has a message board through which the participant could communicate with research therapists (clinical psychologists) who also check completed activities and respond with personalized but standardized messages. Finally, a series of fact sheets cover a range of related topics, including managing SI, plus downloadable relaxation MP3s.

The face-to-face component: Traineed psychologysts will deliver four psychotherapeutic CBT-based sessions (45-min), designed during the formative work (year 1). These sessions will be conducted by school psychologists previously trained, and will help the students in three aspects: i) close support and monitoring in case of an increase of symptomatology; ii) motivation to persist with the intervention; and iii) support the interaction between the students and CBT. The final aim of the inclusion of this component is to maximize the effectiveness of CBT. Two clinical psychologists will supervise the school psychologists (each supervisor will be in charge of 5 schools).

6.1. Control group. Students will receive the Treatment-As-Usual (TAU). It consists of identification and assisted referral to a primary care clinic where trained psychologists will assess the symptomatology and propose a course of actions, from initiation of psychotherapy to referral to a General practitioner to initiate medication if needed.

ELIGIBILITY:
Inclusion Criteria:

* Secondary students aged 13-18 years
* High scores in suicidal ideation, last month (score > 3 in the Columbia Suicide Severity Rating Scale (C-SSRS; Posner et al., 2011)
* Fluent in Spanish language

Exclusion Criteria:

* Suicide attempt(s), last month
* Severe depressive symptoms, assessed by the PHQ-9 (> 3 points)
* High severity of psychotic symptoms assessd by the Community Assessment of Psychic Positive-scale (CAPE, P15, Capra et al., 2013) (cut-off= 1.47, as suggested by Bukenaite et al., 2017)

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 240 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Suicide ideation | One month
  The Suicidal Ideation Questionnaire (SIQ; Reynolds, 1988), a 15-item self-report measure designed to assess suicidal ideation in adolescents. Answers to each item are on a scale from 1 to 7. The scores to each item are summed to generate a total score with a range between 7 and 105. A higher score means higher intensity of suicidal ideation

SECONDARY OUTCOMES:
Suicide attempt | One month
  Two questions assesing whether participants had attempted suicide; if yes, how many attempts
Depressive symptoms | One month
  The adolescent version of the Beck Depression Inventory II (BDI-II; Beck, 1996), is a 21-item scale assessing depresive symtpoms experienced over last two weeks. Answers to each item are on a scale from 0 to 3. The scores to each item are summed to generate a total score with a range between 0 and 63. A higher score means higher intensity of depressive symptoms
Anxiety as trait | One Month
  The State-trait Anxiety Inventory (STAI-X) (Spielberger, Gorsuch & Lushene, 1970), is a self-report questoinnaire with two scales of 20 items each assessing state and trait levels of anxiety. In Trait subscale (STAI-T) respondents indicate how they generally feel on a four point Likert scales from 0 (Almost never) to 3 (Almost always). The minimum score is 0 and the maximum score is 60. A higher score means higher anxiety levels
Anxiety as state | One month
  The State-trait Anxiety Inventory (STAI-X) (Spielberger, Gorsuch & Lushene, 1970), is a self-report questoinnaire with two scales of 20 items each assessing state and trait levels of anxiety. In State subscale (STAI-S) repondents indicate how they generally feel on a four point Likert scales from 0 (Almost never‖) to 3 (Almost always). The minimum score is 0 and the maximum score is 60. A higher score means higher state anxiety levels
Hopelessness | One month
  The Beck Hopelessness Scale (Beck, 1988), is a self-report scale with 20 true or false items, 9 or which are keyed 'false' and 11 are keyed 'true'. For every statement, each response is assigned a score of 0 or 1, and the total hopelessness score is the sum of the scores on the individual items. The minimum score is 0 and the maximum score is 20. A higher score means higher hopelessness levels
Social problem solving | One month
  The Short Form of the Social Problem-Solving Inventory Revised (SPSI-R Short Form) (D'Zurilla et al., 1998). This is a 25-item self-report instrument measuring two adaptive problem-solving dimensions (positive problem orientation and rational problem solving) and three dysfunctional dimensions (negative problem orientation, impulsivity/carelessness style, and avoidance style). Each item is rated on a 5-point scale ranging from not at all true of me (0) to extremely true of me (4). The minimum score is 0 and the maximum score is 75. A higher score means higher social problem solving capability.
Cognitive-behavioral skills | One month
  The Cognitive-Behavioural Therapy Skills Questionnaire (CBTS; Jacob et al., 2011) is a 16-item scale with two scales mesuring two skills: cognitive restructuring (CR) and behavioural activation (BA) (i.e. changes in avoidance/ behavioural control and changes in cognitive style). Respondents rank each item on a 5-point Likert scale from 1 (I don't do this) to 5 (I always do this). The minimum score is 15 and the maximum score is 80. A higher score means higher presence of cognitive-behavioral skills.
Emotional regulation | One month
  The Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA; Gullone &Taffe, 2012) is a 10-item self-report scale assessing two ER styles: Cognitive Reappraisal (CR, 6 items), which consists on redefining a potential emotion-eliciting situation in such a way that its emotional impact is changed; Expressive Suppression (ES, 4 items), which consists on the inhibition of ongoing emotion-expressive behavior. Items are rated 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5). The minimum score is 10 and the maximum score is 50. A higher score means higher presence of emotional regulation styles.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Nuñez, PhD, Principal Investigator — University of Talca
Locations (1):
- Daniel Núñez, Talca, Maule Region, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reynolds, W.M. (1988). Suicidal Ideation Questionnaire: Professional manual. Odessa, FL: Psychological Assessment Resources.
- [Background] Beck, A.T., Steer. R.A., Brown. G.K. (1996) Manual for Beck Depression Inventory-II (BDI-II). San Antonio: The Psychological Corporation.
- [Background] Spielberger, C, Gorsuch, R. & Lushene, R. (1970). Manual for the State-Trait Anxiety Inventory. Palo Alto, California, Consulting Psychologist Press. (Adapt. Española, TEA, 1982).
- [Background] D'Zurilla, T. J., Nezu, A. M., & Maydeu-Olivares, A. (1998). Manual for the social problem-solving inventory-revised. North Tonawanda, New York: Multi-Health Systems
- [Background] Jacob KL, Christopher MS, Neuhaus EC. Development and validation of the cognitive-behavioral therapy skills questionnaire. Behav Modif. 2011 Nov;35(6):595-618. doi: 10.1177/0145445511419254. Epub 2011 Sep 5. PMID 21893554
- [Background] Gullone E, Taffe J. The Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA): a psychometric evaluation. Psychol Assess. 2012 Jun;24(2):409-17. doi: 10.1037/a0025777. Epub 2011 Oct 24. PMID 22023559
- [Background] Capra C, Kavanagh DJ, Hides L, Scott J. Brief screening for psychosis-like experiences. Schizophr Res. 2013 Sep;149(1-3):104-7. doi: 10.1016/j.schres.2013.05.020. Epub 2013 Jul 3. PMID 23830544
- [Background] Bukenaite A, Stochl J, Mossaheb N, Schafer MR, Klier CM, Becker J, Schloegelhofer M, Papageorgiou K, Montejo AL, Russo DA, Jones PB, Perez J, Amminger GP. Usefulness of the CAPE-P15 for detecting people at ultra-high risk for psychosis: Psychometric properties and cut-off values. Schizophr Res. 2017 Nov;189:69-74. doi: 10.1016/j.schres.2017.02.017. Epub 2017 Feb 27. PMID 28254243
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Robinson J, Hetrick S, Cox G, Bendall S, Yung A, Pirkis J. The safety and acceptability of delivering an online intervention to secondary students at risk of suicide: findings from a pilot study. Early Interv Psychiatry. 2015 Dec;9(6):498-506. doi: 10.1111/eip.12136. Epub 2014 Mar 31. PMID 24684927
- [Background] Hetrick SE, Yuen HP, Bailey E, Cox GR, Templer K, Rice SM, Bendall S, Robinson J. Internet-based cognitive behavioural therapy for young people with suicide-related behaviour (Reframe-IT): a randomised controlled trial. Evid Based Ment Health. 2017 Aug;20(3):76-82. doi: 10.1136/eb-2017-102719. Epub 2017 Jul 12. PMID 28701336
- [Derived] Nunez D, Meza D, Andaur J, Robinson J, Gaete J. Reframe-IT+, an indicated preventive school-based intervention, reduces suicidal ideation among adolescents in vulnerable contexts in Chile. BMC Psychol. 2024 Dec 24;12(1):780. doi: 10.1186/s40359-024-02300-9. PMID 39719648